CLINICAL TRIAL: NCT04483986
Title: The Evaluation of Rectus Re-approximation in Terms of Adhesion After Cesarean Section by Elastography.
Brief Title: Does Rectus Re-approximation Cause Adhesion After Cesarean Section?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Giresun University (Other)
Responsible Party: Principal Investigator, Sebnem Alanya Tosun, Assistant Professor, Giresun University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Rectus-reapproximation
Record Dates: First submitted 2020-06-18; First posted 2020-07-23 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Obstetric Complication; Muscle Injury
Keywords: elastography; rectus muscle re-approximation

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Radiologist is blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Active Comparator): This arm is going to include the patients who are performed rectus reapproximation.
  Interventions: Procedure: Rectus muscle re-approximation
- Control group (No Intervention): This arm is going to include the patients who are not performed rectus reapproximation.

INTERVENTIONS:
Procedure: Rectus muscle re-approximation — Study group: we are going to re-approximate rectus muscle wirth minimum 3 stiches.
  Arms: Study group

SUMMARY:
Rectus re-approximation and periton closure are not the obligatory steps during cesarean section. These steps are due to surgeon's preference. However, there is lack of knowledge about the relation of rectus muscle re-approximation and adhesion formation. We are going to study the rectus muscle stiffness by share-wave elastosonography.

ELIGIBILITY:
Inclusion Criteria:

* Primary cesarean section

Exclusion Criteria:

* Wound infection

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2020-05-25 (Actual); Primary Completion 2021-08-25 (Estimated); Study Completion 2021-09-25 (Estimated)

PRIMARY OUTCOMES:
Rectus muscle stiffness | 3 months after cesarean section
  Share wave elastosonography is going to perform to six different points of rectus muscle. Each points will be 2 cm right or left side of linea alba line in horizontal axis. Two points are on cesarean section incision, next two points 2 cm below the incision and other next two points 2 cm above the incision in vertical axis. Rectus muscle stiffness will show the adhesion formation.

SECONDARY OUTCOMES:
Operation time | During operation
  Operation time in minutes is going to be recorded
Postoperative pain | 3 months after cesarean section
  VAS scale is going to be used.
Postoperative bowel function | 3 months after cesarean section
  It is going to be evaluated by self developed questionnaire.
Postoperative bladder function | 3 months after cesarean section
  It is going to be evaluated by self developed questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Sebnem Alanya Tosun, Giresun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No